CLINICAL TRIAL: NCT06160570
Title: Evaluation of Preoperative Chemoradiotherapy Utilizing Intensity Modulated Radiation Therapy (IMRT) When Compared With 3D Conformal Radiotherapy (3DCRT) for Patients With Locally Advanced Rectal Cancer, Prospective Phase II Study.
Brief Title: IMRT Versus 3DCRT for Locally Advanced Rectal Cancer, Prospective Phase II Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMRT versus 3D to rectum
Record Dates: First submitted 2021-02-06; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2021-01

CONDITIONS: Rectal Cancer; Radiotherapy; Toxicity Due to Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT (Active Comparator): Intensive Modulated Radiation Therapy
  Interventions: Radiation: Intensive Modulated Radiation Therapy
- 3DCRT (Active Comparator): 3-Dimension Conformal Radiation Therapy
  Interventions: Radiation: 3-Dimension Conformal Radiation Therapy

INTERVENTIONS:
Radiation: Intensive Modulated Radiation Therapy — Radiotherapy technique: IMRT
  Arms: IMRT
Radiation: 3-Dimension Conformal Radiation Therapy — Radiotherapy technique: 3DCRT
  Arms: 3DCRT

SUMMARY:
The goal of this prospective phase II study was to determine whether personalized planning-based nCRT for LARC would indeed decrease small bowel dose, and whether selected plans, specifically prioritizing lower dose to small bowel, would result in lower rates of acute GI toxicity compared with previously reported rates.

DETAILED DESCRIPTION:
The standard of care for locally advanced rectal cancer is neoadjuvant chemoradiotherapy. However, acute gastrointestinal (GI) toxicity is common. Some retrospective studies suggested that Intensity Modulated Radiation Therapy( IMRT) reduces acute bowel toxicity compere to 3D conformal radiotherapy (3DCRT).The aim of this prospective phase II study to determine whether the use of IMRT planning in neoadjuvant chemoradiotherapy in patients with locally advanced rectal cancer can decrease small bowel irradiation dose compared to commonly used 3D conformal techniques ,and the rate of acute GI toxicity.

Patients (pts) with clinical stage II-III rectal adenocarcinoma were enrolled in a prospective phase II study of preoperative chemoradiation. For each patient two radiation plans were performed: IMRT and 3DCRT. After comparing two DVH (dose volume histogram) plans for organs at risk (OARs), such as small bowel and bladder, pts were treated according to the plan with maximal critical organs sparing. All Patients received 45 Gy in 25 fractions to the rectum and draining lymph nodes, followed by boost to the tumor, with concurrent capecitabine or 5- Fluorouracil .Weekly follow up was performed to assess acute toxicity.

The investigators hypothesize that the use of IMRT in neoadjuvant chemoradiation for locally advanced rectal cancer may reduce the small bowel and bladder irradiated volume and consequently reduce acute toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced rectal adenocarcinoma
* Performance status of 0-2
* Adequate hematologic, renal, and hepatic function

Exclusion Criteria:

* Prior radiotherapy to pelvis
* Metastatic disease at diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related gastrointestinal and urinary adverse events as assessed by CTCAE v5.0 | 3 months
  Acute gastrointestinal and urinary toxicity

SECONDARY OUTCOMES:
Pathological response to chemoradiotherapy | 3 months
  Pathological response to neoadjuvant chemoradiotherapy was assessed on the surgical specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Kundel, MD, Principal Investigator — Davidoff Cancer Center, Rabin Medical Center
Locations (1):
- Orly Yariv, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No